## TRANSLATION FROM SWEDISH MAY 29 2018

Visualization of Asymptomatic Atherosclerotic Disease for Optimum Cardiovascular Prevention: VIPVIZA – a Population-based RCT nested in Routine Care in Sweden

NCT01849575

Informed consent, translation from Swedish to English

## TRANSLATION FROM SWEDISH MAY 29 2018



| Informed consent | Personal id number |
|---|---|
| I hereby certify that I have received oral and writte<br>requirement for an ultrasound examination of the<br>join the trial when I participated in the Västerbotte | neck (carotid) arteries, and that I was invited to |
| ☐ <b>YES</b> I consent to participate in the study and will randomly be allocated to informed or not infor examination. I am also aware that individuals who not be included in the study but will be offered a re Hospital. I am also aware that among trial participathe neck arteries, a smaller group will receive more monitoring. | med about the results of the ultrasound have severe stenosis of the carotid arteries will eferral to the Stroke Center, Umeå University ants who have moderately pronounced changes in |
| I am also aware that my participation is complewithout further explanation, I can withdraw more within the healthcare system. | |
| I consent to the authorized representative(s) of this with the above information, including data in my metal pharmacological prescription, and cardiovascular description of information from the Pharmacological Welfare regarding purchase of prescribed pharmacological diseases during the same period, as surgical procedures, myocardial infarctions and streat the National Board of Health and Welfare. | nedical records on cardiovascular risk factors,<br>lisease events for 10 years. I also consent to<br>Registry at the National Board of Health and<br>cological treatments aiming at prevention of<br>well as retrieval of data on revascularizating |
| I consent to this, provided there is full confider | ntiality during handling of the data. |
| <u>Please sign below</u> and also write your address, you, including during office hours | email and phone number so we can reach |
| □ <b>NO</b> I do not consent to participate in this | study <u>Please sign below</u> |
| Place Date/20 | Signature |
| Printe | d name |
| Nurse: I have given oral and written information | on about the study to the above person: |
| Place Date/20 | Signature |
| Health care center Print | ed name |

## TRANSLATION FROM SWEDISH MAY 29 2018

## If you answered YES: Contact information:

| Address |
|--------------------------------------------------------------|
| Mail address |
| Phone number |
| Mobile number |
| ☐ Lagree to get a reminder with SMS prior to the study visit |